CLINICAL TRIAL: NCT01187173
Title: The Fibrosis-Lymphedema Continuum in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sheila Ridner, Professor, Vanderbilt University
Other Study IDs: 100475
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Neoplasms; Fibrosis; Lymphedema; Biomarkers; Polymorphism, Genetic; Depression
MeSH Terms: conditions — Head and Neck Neoplasms; Fibrosis; Lymphedema; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood from blood draws
Oversight: Data Monitoring Committee: No

SUMMARY:
Goal:

The primary goal of this study is to longitudinally investigate, in head and neck cancer (HNC) patients, the potential fibrosis-lymphedema continuum. Specifically, we will examine the development, patterns, progression, and prevalence of late-effect fibrosis and/or lymphedema, explore potential biological correlatives including pro-inflammatory cytokines and genetic polymorphisms, and evaluate the relationship among late-effect fibrosis and/or lymphedema and select psychosocial stressors that potentially interact with cytokine pathways.

H: A minimum of 20 percent of HNC patients will experience late-effect fibrosis and/or lymphedema.

H: We will be able to differentiate characteristics patterns of the development of late-effect fibrosis and/or lymphedema.

H: We will be able to differentiate patterns of symptoms associated with late-effect fibrosis and/or lymphedema.

H: We will be able to differentiate patterns of inflammatory response and the development of late-effect fibrosis and/or lymphedema.

H: Select polymorphisms will increase the likelihood of development of late-effect fibrosis and/or lymphedema.

H: Incidence and severity of late-effect fibrosis and/or lymphedema will correlate with total dose of radiation to involved anatomical site.

H: HNC patients with fibrosis and/or lymphedema experience greater levels of depression and social withdrawal than those without these conditions.

DETAILED DESCRIPTION:
Background: The use of aggressive treatment for HNC, particularly combined modality treatment regimens has resulted in an increase in survival. Unfortunately, this improvement has come with a marked increase in acute and late-effects. These undesirable treatment outcomes exact a heavy toll on functional capacity, contribute to a myriad of problematic physical and psychological symptoms, negatively impact Quality of Life, and likely create a significant economic burden to both the patients and the health care system.

Objective: This four year, longitudinal study will examine the development, patterns, nature, progression, and prevalence of late-effect fibrosis and/or lymphedema, explore potential host biological correlatives (pro-inflammatory cytokines and genetic polymorphisms), and examine select psychological stressors (depression, social withdrawal), associated with late-effect fibrosis and lymphedema in HNC survivors.

Specific Aims:1. To determine the prevalence and nature of late-effect (≥3 months post-treatment) fibrosis and/or lymphedema in HNC patients. 2. To explore the relationships among the biological mechanisms of inflammatory response, genetic polymorphisms, treatment factors, and late-effect fibrosis and/or lymphedema in HNC patients. 3. To explore the relationships among late-effect fibrosis and/or lymphedema and psychosocial stressors (depression and social withdrawal) in HNC patients.

Study Design: HNC patients will be assessed at baseline, end of treatment (EOT), and every six weeks after treatment up to one year after treatment, and twice more at 15 and 18 months post-treatment. These intervals were chosen to reduce subject burden as they routinely coincide with scheduled laryngoscopic procedures. At baseline, the follow assessment will be undertaken: 1) demographic information and alcohol and tobacco use history; 2) disease characteristics; 3) presence of tumor related fibrosis and/or lymphedema (laryngoscope with digital photographs and scoring of internal lymphedema with Patterson Scale) and external fibrosis/lymphedema with digital photography, physical exam for fibrosis/lymphedema using the Foldi criteria, and CT scans; 4) blood for inflammatory mediators and polymorphisms; 5) psychosocial assessments (Center for epidemiological Studies Depression Scale, Liebowitz Anxiety Scale); and 6) functional assessments (MBVS, Cervical Range of Motion [CROM], Neck Disability Index and VHNSS). Post-treatment, and every scheduled assessment thereafter, patients will undergo repeat assessments for everything except: demographic information, medical history, ETOH and smoking history, polymorphisms and MBVs.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed, histologically proven carcinoma involving the head and neck
* Stage II or greater
* age of 21 or over
* willing and able to undergo baseline and follow-up assessment at the VICC Nashville, or the Nashville Veterans Administration Medical Center (Nashville VA
* the ability to speak English

Exclusion Criteria:

* medical record documentation of cognitive impairment that would preclude the ability to provide informed consent
* unwilling to undergo routine follow-up at VICC Nashville or the Nashville VA
* recurrent cancer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population consists of patients with carcinoma of the head and neck. Subjects will be recruited from newly diagnosed patients with carcinoma of the head and neck undergoing treatment at the VICC, Vanderbilt Cool Springs Clinic, and the Nashville Veterans Administration (VA) Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Prevelence and nature of fibrosis and/or lymphedema | baseline, every six wks. first year pot-tx, and 15 & 18 mths post tx.
Relationships among biological mechanisms of fibrosis and/or lymphedema | baseline, every 6 weeks after tx. for one year, and 15 and 18 months after tx.
Relationship of fibrosis and/or lymphedema and psychosocial stressors | baseline, every 6 weeks post tx for 1 year and 15 and 18 months post tx.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Ingram Cancer Center, Nashville, Tennessee, United States